CLINICAL TRIAL: NCT02953262
Title: Improving Diabetes Care Through Effective Personalized Patient Portal Interactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-307
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Personal Health Records; Patient Outcome Assessment; Mental Health
MeSH Terms: conditions — Diabetes Mellitus; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not explicitly told which group they were randomized to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Encouragement Arm 1 (Experimental): Participants in this encouragement condition will receive a mailed brochure with basic My HealtheVet content and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
  Interventions: Behavioral: My HealtheVet Brochure; Behavioral: My HealtheVet Training Guide for Veterans Living with Diabetes; Behavioral: My HealtheVet Group Training; Behavioral: My HealtheVet Individual Training
- Encouragement Arm 2 (Experimental): Participants in this encouragement condition will receive the same brochure and training guide as Arm 1 but will also be offered optional attendance at one of several group training sessions.
  Interventions: Behavioral: My HealtheVet Brochure; Behavioral: My HealtheVet Training Guide for Veterans Living with Diabetes; Behavioral: My HealtheVet Group Training
- Encouragement Arm 3 (Experimental): Participants in this encouragement condition will receive the same as in Arm 2 (brochure, training guide, and group training offer) but will also be offered a one-on-one My HealtheVet training session.
  Interventions: Behavioral: My HealtheVet Training Guide for Veterans Living with Diabetes; Behavioral: My HealtheVet Group Training
- Brochure Only Comparison Arm (Other): The Comparison condition will only receive a mailed brochure with basic My HealtheVet content during the trial. (The training guide will be mailed to them after completion of the interview at the end.)
  Interventions: Behavioral: My HealtheVet Group Training

INTERVENTIONS:
Behavioral: My HealtheVet Brochure — Participants will receive a mailed brochure with basic My HealtheVet content.
  Arms: Encouragement Arm 1; Encouragement Arm 2
Behavioral: My HealtheVet Training Guide for Veterans Living with Diabetes — Participants will be mailed a bound My HealtheVet training guide with step by step instructions on how to register, upgrade to Premium account, refill prescriptions, use secure messaging, download their Blue Button reports, and other features
  Arms: Encouragement Arm 1; Encouragement Arm 2; Encouragement Arm 3
Behavioral: My HealtheVet Group Training — Participants will be invited to participate in a scheduled group training to learn how to use My HealtheVet to help manage their diabetes
Behavioral: My HealtheVet Individual Training — Participants will be invited to participate in a one-on-one training to learn how to use My HealtheVet to help manage their diabetes at a time of their convenience.
  Arms: Encouragement Arm 1

SUMMARY:
Patient-facing eHealth technologies, such as online patient portals, connect patients with the healthcare system, help them access their health information, and support self-management of health conditions. This study tested an intervention to improve adoption and use of the My HealtheVet patient portal for diabetes management.

DETAILED DESCRIPTION:
The goal of this small scale study is to test the feasibility of engaging Veterans in a supported adoption intervention to promote effective patient portal use in a sample of Veterans with uncontrolled Type II diabetes.

Participants were eligible for recruitment if they were Veterans age 18-85 who were actively receiving care at one of the study sites (as determined by having an upcoming scheduled appointment), had uncontrolled glucose (HbA1c >= 8.5%), and had either never used the VA patient portal or were inactive registrants who have not used the patient portal in the past 12 months. Participants who met these conditions and did not opt out of the study were randomized to one of four arms: 1) Encouragement I (brochure + mailed training guide), 2) Encouragement II (brochure + mailed training guide + invitation to group training), 3) Encouragement III (brochure + mailed training guide + invitation to group and one-on-one training), and 4) Comparison (standard patient portal enrollment brochure only). All arms received the standard My HealtheVet patient portal enrollment brochure along with an invitation to participate in the study. Those randomized to any of the Encouragement Arms received a mailed training guide. The My HealtheVet Training Guide for Veterans Living with Diabetes was designed in conjunction with Veteran co-investigators based on feedback from patients living with diabetes who were My HealtheVet users. It provided step by step guidance on how to use the features Veterans living with diabetes find most helpful with specific examples of use for diabetes self-management. Those in Encouragement Arm II were also invited to attend one of several group training sessions. Those in Encouragement III were invited to schedule a one-on one session to learn how to use the patient portal. Those in the comparison condition were asked during their interview if they would like a Training Guide mailed to them at the end of the trial, and those interested were mailed a Training Guide.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Hemoglobin A1c result >=8.5% at most recent lab test prior to recruitment
* Non use of the VA patient portal, defined by not being registered or registered with no activity in 12 months
* Currently being seen at one of the sites participating in the study (upcoming appointment scheduled)

Exclusion Criteria:

* Non-Veterans
* Controlled hemoglobin A1c levels (A1c<8.5%) at most recent lab test prior to recruitment
* Recent use of the patient portal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Shimada, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (2):
- United States (2):
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robinson SA, Zocchi MS, Netherton D, Ash A, Purington CM, Connolly SL, Vimalananda VG, Hogan TP, Shimada SL. Secure Messaging, Diabetes Self-management, and the Importance of Patient Autonomy: a Mixed Methods Study. J Gen Intern Med. 2020 Oct;35(10):2955-2962. doi: 10.1007/s11606-020-05834-x. Epub 2020 May 21. PMID 32440998
- [Result] Stewart MT, Hogan TP, Nicklas J, Robinson SA, Purington CM, Miller CJ, Vimalananda VG, Connolly SL, Wolfe HL, Nazi KM, Netherton D, Shimada SL. The Promise of Patient Portals for Individuals Living With Chronic Illness: Qualitative Study Identifying Pathways of Patient Engagement. J Med Internet Res. 2020 Jul 17;22(7):e17744. doi: 10.2196/17744. PMID 32706679
- [Result] Zocchi MS, Robinson SA, Ash AS, Vimalananda VG, Wolfe HL, Hogan TP, Connolly SL, Stewart MT, Am L, Netherton D, Shimada SL. Patient portal engagement and diabetes management among new portal users in the Veterans Health Administration. J Am Med Inform Assoc. 2021 Sep 18;28(10):2176-2183. doi: 10.1093/jamia/ocab115. PMID 34339500
- [Result] Robinson SA, Netherton D, Zocchi M, Purington C, Ash AS, Shimada SL. Differences in Secure Messaging, Self-management, and Glycemic Control Between Rural and Urban Patients: Secondary Data Analysis. JMIR Diabetes. 2021 Nov 19;6(4):e32320. doi: 10.2196/32320. PMID 34807834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting eligibility criteria were identified from clinical records and mailed an invitation to participate in the study along with a My HealtheVet brochure and an information sheet describing the study. Initial invitations were sent out in June 2019 at Site 1 and in December 2019 at Site 2. Patients who did not opt out were enrolled and randomized into study arms in July 2019 and January 2020, respectively.
Pre-assignment Details: One patient was mistakenly randomized to an arm even though he was deceased shortly prior to enrollment because he met the eligibility criteria according to our databases, including having a future appointment scheduled. Fifteen patients from one site were incorrectly identified as not having used the portal in the 12 months prior to the trial and were excluded from the analyses.
Groups:
- Brochure Only Comparison Arm: The comparison condition only received a mailed brochure with basic My HealtheVet content during the trial.
  After the completion of their interview, they were offered a copy of the training guide.
- Encouragement Arm 1: Participants in this encouragement condition received a brochure about the My HealtheVet portal and were mailed a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
- Encouragement Arm 2: Participants in this encouragement condition received the My HealtheVet brochure and training guide, but was also offered optional attendance at one of several group training sessions.
- Encouragement Arm 3: Participants in this encouragement condition received the same encouragement as in Arm 2 (brochure, training guide and group training offer) but were also offered a one-on-one My HealtheVet training session.
Period: Overall Study
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
Started | 68 | 69 | 68 | 70
Completed | 65 | 63 | 65 | 67
Not Completed | 3 | 6 | 3 | 3
Not completed — Used portal during 6 months prior to randomization | 3 | 6 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Brochure Only Comparison Arm: The comparison condition only received a mailed brochure with basic My HealtheVet content during the trial.
  After the completion of their telephone interview, they were offered a copy of the training guide.
- Encouragement Arm 1: Participants in this encouragement condition received a brochure about the My HealtheVet portal and were also mailed a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
- Encouragement Arm 2: Participants in this encouragement condition received the My HealtheVet brochure and training guide, but were also offered optional attendance at one of several group training sessions.
- Total: Total of all reporting groups
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3 | Total
Number analyzed (Participants) | 65 | 63 | 65 | 67 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10.3) | 68.3 (8.8) | 68.5 (8.8) | 70.0 (9.1) | 68.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 0 | 5
  Male | 63 | 62 | 63 | 67 | 255
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 54 | 47 | 57 | 55 | 213
  Black/African-American | 5 | 6 | 4 | 5 | 20
  Latino | 4 | 5 | 4 | 0 | 13
  Other | 0 | 1 | 0 | 2 | 3
  Unknown/Missing | 2 | 4 | 0 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 63 | 65 | 67 | 260
Rural Residence [Count of Participants; unit: Participants] | 0 | 2 | 3 | 2 | 7
Marital Status [Count of Participants; unit: Participants]
  Married | 30 | 30 | 31 | 34 | 125
  Widowed | 4 | 4 | 5 | 3 | 16
  Divorced/Separated | 19 | 14 | 24 | 18 | 75
  Single | 12 | 15 | 5 | 12 | 44
Average HbA1c at baseline (2019) [Mean (Standard Deviation); unit: % (DCCT units)] | 9.6 (1.3) | 9.3 (1.0) | 9.5 (1.3) | 9.3 (1.1) | 9.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Any My HealtheVet Patient Portal Use
Description: This measure captures any use of MHV within 180 days of the brochure mailing, including use of prescription refills, secure messaging, Blue Button, or any other portal features.
Time Frame: Portal use within 180 days of initial brochure mailing
Population: Patients randomized to each arm who had not used My HealtheVet in the 12 months prior to randomization. At the second site, 15 people who should have been excluded were inadvertently included in the sample because the criteria of no secure messaging use in previous 12 months was mistakenly used instead of no patient portal use in the previous 12 months. We did not discover this until after the trial was complete because there were delays in receiving actual portal use data.
Measure: Count of Participants; unit: Participants
Groups:
- Brochure Only Comparison Arm: The Comparison condition will only receive a mailed brochure with basic My HealtheVet content during the trial. (The training guide will be mailed to them after completion of the 6-month interview.)
  Brochure Only Intervention 4: Participants will receive a mailed brochure with basic My HealtheVet content.
- Encouragement Arm 1: Participants in this encouragement condition will receive a mailed brochure with basic My HealtheVet content and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
  Supported Adopted Intervention 1: Participants in this encouragement condition will receive a mailed brochure and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
  Brochure Only Intervention 4: Participants will receive a mailed brochure with basic My HealtheVet content.
- Encouragement Arm 2: Participants in this encouragement condition will receive the same brochure and training guide as Arm 1 but will also be offered optional attendance at one of several group training sessions.
  Supported Adopted Intervention 1: Participants in this encouragement condition will receive a mailed brochure and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
  Supported Adopted Intervention 2: Participants will be offered optional attendance at a group training session in addition to receiving the brochure and training guide by mail. These sessions will be offered at a computer lab at the VA hospital.
  Brochure Only Intervention 4: Participants will receive a mailed brochure with basic My HealtheVet content.
- Encouragement Arm 3: Participants in this encouragement condition will receive the same as in Arm 2 (brochure, training guide, and group training offer) but will also be offered a one-on-one My HealtheVet training session.
  Supported Adopted Intervention 1: Participants in this encouragement condition will receive a mailed brochure and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
  Supported Adopted Intervention 2: Participants will be offered optional attendance at a group training session in addition to receiving the brochure and training guide by mail. These sessions will be offered at a computer lab at the VA hospital.
  Supported Adopted Intervention 3: Participants will also be offered a one-on-one My HealtheVet training session in addition to the brochure, training guide, and offer of group training session.
  Brochure Only Intervention 4: Participants will receive a mailed brochure with basic My HealtheVet content.
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
Number analyzed (Participants) | 65 | 63 | 65 | 67
Participants | 6 | 1 | 5 | 8
Statistical Analysis 1: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 1; Test type: Superiority; p = 0.057, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 2; Test type: Superiority; p = 0.753, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 3; Test type: Superiority; p = 0.613, Chi-squared — The a priori threshold for statistical significance was p=0.05

2. Secondary Outcome: Patient Upgraded to a Premium My HealtheVet Portal Account
Description: After registering for the portal, patients must confirm their identity and accept the terms and conditions of the portal in order to upgrade to Premium status which allows access to secure messaging, their VA appointments, and electronic health record extracts such as lab results, medical imaging and reports, clinical notes, and their VA health summary. Patients can access a limited subset of portal features, including online prescription refills, without upgrading to Premium. This measure captures whether a participant upgraded to a Premium account during the trial.
Time Frame: 180 days from brochure mailing
Measure: Count of Participants; unit: Participants
Groups:
- Brochure Only Comparison Arm: The Comparison condition will only receive a mailed brochure with basic My HealtheVet content during the trial. (The training guide will be mailed to them after completion of the interview at the end.)
  My HealtheVet Brochure: Participants will receive a mailed brochure with basic My HealtheVet content.
- Encouragement Arm 3: Participants in this encouragement condition will receive the same as in Arm 2 (brochure, training guide, and group training offer) but will also be offered a one-on-one My HealtheVet training session.
  My HealtheVet Brochure: Participants will receive a mailed brochure with basic My HealtheVet content.
  My HealtheVet Training Guide for Veterans Living with Diabetes: Participants will be mailed a bound My HealtheVet training guide with step by step instructions on how to register, upgrade to Premium account, refill prescriptions, use secure messaging, download their Blue Button reports, and other features
  My HealtheVet Group Training: Participants will be invited to participate in a scheduled group training to learn how to use My HealtheVet to help manage their diabetes
  My HealtheVet Individual Training: Participants will be invited to participate in a one-on-one training to learn how to use My HealtheVet to help manage their diabetes at a time of their convenience.
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
Number analyzed (Participants) | 65 | 63 | 65 | 67
Participants | 0 | 1 | 2 | 5
Statistical Analysis 1: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 1; Test type: Superiority; p = 0.308, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 2; Test type: Superiority; p = 0.154, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 3; Test type: Superiority; p = 0.025, Chi-squared — The a priori threshold for statistical significance was p=0.05

3. Secondary Outcome: Use of Online Prescription Refills
Description: This measure captures whether the participant used the portal's online prescription refill feature at least once within 180 days of mailing the brochure.
Time Frame: 180 days from brochure mailing
Measure: Count of Participants; unit: Participants
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
Number analyzed (Participants) | 65 | 63 | 65 | 67
Participants | 5 | 1 | 0 | 3
Statistical Analysis 1: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 1; Test type: Superiority; p = 0.102, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 2; Test type: Superiority; p = 0.023, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 3; Test type: Superiority; p = 0.439, Chi-squared — The a priori threshold for statistical significance was p=0.05

4. Secondary Outcome: Use of Secure Messaging
Description: Patient used the secure messaging feature during the trial
Time Frame: 180 days from brochure mailing
Measure: Count of Participants; unit: Participants
Arm/Group | Brochure Only Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
Number analyzed (Participants) | 65 | 63 | 65 | 67
Participants | 1 | 1 | 2 | 7
Statistical Analysis 1: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 1; Test type: Superiority; p = 0.982, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 2; Test type: Superiority; p = 0.559, Chi-squared — The a priori threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Brochure Only Comparison Arm vs Encouragement Arm 3; Test type: Superiority; p = 0.032, Chi-squared — The a priori threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 180 days for each participant
Description: Patient deaths during the trial were typically discovered from communication with family members when reaching out to participants by telephone to schedule a training session or interview. These deaths were unrelated to participation in the trial but were reported to the institutional review board when discovered.
Groups:
- Comparison Arm: The Comparison condition received a mailed brochure with basic My HealtheVet information.
  They were offered a training guide at the end of the study (after their interview).
- Encouragement Arm 1: Participants in this encouragement condition received the mailed brochure and a training guide with (a) insights from other Veterans on how to use My HealtheVet for diabetes self-management, (b) step-by-step guidance for how to sign up for My HealtheVet and, (c) detailed guidance on how to learn to use key features.
- Encouragement Arm 2: Participants in this encouragement condition received the brochure and the same training guide as Arm 1 but were also offered optional attendance at one of several group training sessions.
- Encouragement Arm 3: Participants in this encouragement condition received the same as in Arm 2 (brochure, training guide and group training offer) but were also offered a one-on-one My HealtheVet training
Arm/Group | Comparison Arm | Encouragement Arm 1 | Encouragement Arm 2 | Encouragement Arm 3
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/69 | 4/68 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/68 | 0/70
Other Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/68 | 0/70

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, group and one-on-one sessions planned at the second site had to be converted to virtual sessions without a hands-on component. This led to lower participation in training sessions at this second site.

At the second site, 15 people who had portal activity in the previous year were inadvertently included. These 15 people were excluded from analysis of outcomes.

Only a subset of those enrolled in each arm completed the telephone interview.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT02953262/Prot_SAP_000.pdf